CLINICAL TRIAL: NCT06407466
Title: The Effect of Soft Tissue Mobilization and Kinesio Taping Applied to Athletics Athletes on Sports Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar5
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Athletic Injuries; Sports Physical Therapy
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- taping (Experimental): kinesiotape
  Interventions: Other: taping
- mobilization (Experimental): instrument-assisted soft tissue mobilization
  Interventions: Other: mobilization
- control (Active Comparator): Those who did not receive any intervention
  Interventions: Other: Control

INTERVENTIONS:
Other: taping — Kinesiology taping; In order to facilitate the muscle, while the subject is standing and his body is flexed to ensure hip flexion, both "I" bands will be applied from the origin to the insertion, with 30% stretching from the medial and lateral, starting from the Ischial Tuberositas to the border of the Popliteal Fossa.
  Arms: taping
Other: Control — The routine training program will continue without intervention.
  Arms: control
Other: mobilization — Instrument-assisted soft tissue mobilization; The subject is in a prone position on a bed, with the lower extremity in a neutral position, and a hazelnut-sized amount of lubricant will be applied to the working surface, and will be applied to the skin on the back of the upper leg for 5 minutes, targeting the tissue structures. (Hamstring and deep fascia covering this muscle) Pressure and speed will be adjusted according to the subject's tolerance so as not to cause pain.
  Arms: mobilization

SUMMARY:
The aim of the research is to evaluate the effects of tool-assisted soft tissue mobilization and kinesiology tape applications applied to the Hamstring muscle on balance, agility and jumping in athletics athletes.

DETAILED DESCRIPTION:
Participants will be divided into 3 groups. Kinesiology taping will be applied to the 1st group, and instrument-assisted soft tissue mobilization will be applied to the 2nd group. The 3rd group will be the control group and no application will be made. All 3 groups will participate in regular training. Before training, applications will be made to the Hamstring muscle on both legs. All 3 groups will be evaluated before, after and 1 month after training, and the 1st and 2nd groups will be evaluated by comparing them with the 3rd group (control group). A 15-minute warm-up period will be given before the measurements. During the post-application measurements, the 1st group will have Kinesiological Taping. There will be 3-minute rest periods between measurements to prevent fatigue. Kinesiology taping; In order to facilitate the muscle, while the subject is standing and his body is flexed to ensure hip flexion, both "I" bands will be applied from the origin to the insertion, with 30% stretching from the medial and lateral, starting from the Ischial Tuberositas to the border of the Popliteal Fossa. Instrument-assisted soft tissue mobilization; The subject is in a prone position on a bed, with the lower extremity in a neutral position, and a hazelnut-sized amount of lubricant will be applied to the working surface, and will be applied to the skin on the back of the upper leg for 5 minutes, targeting the tissue structures. (Hamstring and deep fascia covering this muscle) The pressure and speed will be adjusted according to the tolerance of the subject so as not to cause pain. Participants will be administered the Unipedal Stance Test, Agility T-Test and Standing Long Jump Test.

ELIGIBILITY:
Inclusion criteria

* Have been doing athletics for the last 6 months and participate in training regularly,
* Are between the ages of 10-40,
* Those who train at least 3 days a week,
* Athletes who have consent to participate in the study (athletes between the ages of 10-18 with consent from their parents) will be included.

Exclusion criteria

* Having any history of injury or acute infection,
* Having a systemic and metabolic disease,
* Having a history of chronic pain,
* Having an unhealed or unstable bone fracture,
* Athletes with allergies, infections or open wounds on the skin will not be included.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Unipedal Stance Test | 6 weeks
  It is a static balance test. For the test, participants are asked to stand on their chosen foot; the other foot is lifted (it should be close to but not touching the ankle on the floor), while the arms are positioned diagonally across the chest. You are told to focus on a point at eye level during the test. When the participant lifts his feet off the ground, time calculation begins using a stopwatch. The time calculation ends when the participant does one of the following: Uses arms (i.e. does not cross arms), uses lifted foot, moves weight-bearing foot to maintain balance. The process is repeated 3 times and the best of 3 attempts is recorded. A 5-minute rest is allowed between each set of trials to prevent fatigue.There is no maximum minimum wage.
Agility T Test | 6 weeks
  The T test consists of 4 contact points formed in a T shape in an area of 10m length and 10m width. The aim is to complete a series that requires the subject to move in different directions and in different ways between these contact points in the shortest time possible. The difference between this test and other agility tests is that the subject always looks in the same direction. It changes direction by sliding steps to the right and left or by running backwards. This test requires two 900° and 1800° turns, as well as 10m forward, 10m right, 10m left and 10m back, for a total distance of 40m. The subjects' toes are placed just behind the line, their feet are at normal range, they are parallel to the ground, their arms are in front, their knees are bent, they jump as far as they can with the arms swinging, and both feet touch the ground at the same time. The test is repeated twice and the athletes' best distance is recorded in meters.There is no maximum minimum wage.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu KARACALİOĞLU, Study Chair — Uskudar University
Locations (1):
- Uskudar Üniversity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rana A, Tyagi D, Alghadir AH, Khan M. Effects of Kinesio taping on calf muscle fatigue in college female athletes: A randomized controlled trial. Medicine (Baltimore). 2022 Oct 28;101(43):e31004. doi: 10.1097/MD.0000000000031004. PMID 36316875
- [Background] Ikeda N, Otsuka S, Kawanishi Y, Kawakami Y. Effects of Instrument-assisted Soft Tissue Mobilization on Musculoskeletal Properties. Med Sci Sports Exerc. 2019 Oct;51(10):2166-2172. doi: 10.1249/MSS.0000000000002035. PMID 31083046
- [Background] Kim J, Sung DJ, Lee J. Therapeutic effectiveness of instrument-assisted soft tissue mobilization for soft tissue injury: mechanisms and practical application. J Exerc Rehabil. 2017 Feb 28;13(1):12-22. doi: 10.12965/jer.1732824.412. eCollection 2017 Feb. PMID 28349028
- [Background] Mostafavifar M, Wertz J, Borchers J. A systematic review of the effectiveness of kinesio taping for musculoskeletal injury. Phys Sportsmed. 2012 Nov;40(4):33-40. doi: 10.3810/psm.2012.11.1986. PMID 23306413
- [Background] Kaya Kara O, Atasavun Uysal S, Turker D, Karayazgan S, Gunel MK, Baltaci G. The effects of Kinesio Taping on body functions and activity in unilateral spastic cerebral palsy: a single-blind randomized controlled trial. Dev Med Child Neurol. 2015 Jan;57(1):81-8. doi: 10.1111/dmcn.12583. Epub 2014 Sep 12. PMID 25213082